CLINICAL TRIAL: NCT03867383
Title: Calcium Chloride in the Prevention of Uterine Atony During Cesarean in Women at Increased Risk of Hemorrhage: a Pilot Randomized Controlled Trial and Pharmacokinetic Study
Brief Title: Calcium Chloride for Prevention of Uterine Atony During Cesarean
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 43076
Record Dates: First submitted 2018-04-20; First posted 2019-03-08 (Actual); Results first posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Uterine Atony; Uterine Atony With Hemorrhage; Cesarean Section Complications
MeSH Terms: conditions — Uterine Inertia | interventions — Calcium Chloride; Calcium; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients are randomized via stratified, permuted block randomization to receive a single dose of either calcium chloride 1 gram administered intravenously or placebo at the time of fetal delivery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization has been performed and study ID designation to drug or placebo arm allocated to opaque envelopes prior to subject enrollment. An anesthesiologist not involved in clinical care of the patient or data entry or analysis opens the envelope at the time of subject enrollment and prepares the study drug versus placebo in a 60mL syringe, labeled only with subject ID#. Drug and placebo appear identical as clear solutions and are administered by the same protocol.
  The key designating whether each study ID patient received calcium or placebo has been uploaded to the redCAP data entry database and cannot be retrieved without entering a passcode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium Chloride (Experimental): Non-participating anesthesiologist prepares the drug solution, which is 1 gram of calcium chloride diluted into a total volume of 60 milliliters normal saline, labeled only with the study ID number. The solution is administered intravenously utilizing an Alaris syringe pump and microbore tubing, with infusion starting immediately at the time of fetal delivery at a rate of 360 milliliters per hour (for a calcium infusion rate of 100 milligrams /minute until the full 1 gram dose is administered).
  This is a one-time administration. Patients continue to receive all standard care during the Cesarean including 1 unit oxytocin bolus at the time of fetal delivery + continuous oxytocin infusion at 7.5 units per hour per our institution's protocol.
  Interventions: Drug: Calcium Chloride
- Placebo (Placebo Comparator): Non-participating anesthesiologist prepares the placebo solution, which is 60 milliliters normal saline, labeled only with the study ID number. The solution is administered intravenously utilizing an Alaris syringe pump and microbore tubing, with infusion starting immediately at the time of fetal delivery at a rate of 360 milliliters per hour.
  This is a one-time administration. Patients continue to receive all standard care during the Cesarean including 1 unit oxytocin bolus at the time of fetal delivery + continuous oxytocin infusion at 7.5 units per hour per our institution's protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium Chloride — All included in intervention description.
  1 gram of calcium chloride in total 60 milliliters normal saline
  Other Names: calcium chloride intravenous; IV calcium
  Arms: Calcium Chloride
Drug: Placebo — 60 milliliters normal saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
In this pilot study, investigators will administer calcium chloride or placebo to pregnant women undergoing Cesarean delivery who have been identified as high risk for hemorrhage due to poor uterine muscle contraction, or atony. They will assess whether a single dose of calcium given immediately after the delivery of the fetus decreases the incidence of uterine atony and bleeding for the mother. The pharmacokinetics of calcium chloride in pregnant women will also be established. Data from this pilot study of 40 patients will be used to determine sample size and appropriateness of a larger randomized clinical trial.

DETAILED DESCRIPTION:
Poor contraction of the uterus, also known as uterine atony, is the leading cause of severe blood loss during Cesarean section, both in the US and worldwide. Exogenous calcium has been shown to increase uterine muscle contraction in in vitro and in animal studies. Calcium is also an essential factor in normal blood clotting. Anesthesiologists commonly administer intravenous calcium chloride during Cesarean as well as other types of surgery, but formal randomized studies to determine efficacy in improving uterine tone have not been performed.

In this pilot, randomized controlled study, the anesthesiologist will administer a one-time dose of intravenous calcium chloride 1gram versus placebo at the time of fetal delivery to women identified as having high risk of hemorrhage during Cesarean delivery. Primary outcome assessed will be a composite measure of uterine atony. Data from the pilot study will be used to perform power and sample size calculations for a larger study. Secondary outcomes assessed will include total blood loss, subjective assessment of uterine tone by the blinded obstetrician performing surgery, safety, side effects, and pharmacokinetic profile of calcium chloride in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

Pregnant female subjects at Lucile Packard Children's hospital / Stanford hospital undergoing Cesarean will be screened for inclusion in the study based upon presence of at least 2 risk factors for uterine atony/ postpartum hemorrhage. The risk factors include the following:

* intrapartum Cesarean delivery
* failed operative vaginal delivery with forceps or vacuum
* magnesium infusion
* chorioamnionitis
* multiple gestation
* polyhydramnios
* preterm delivery <37 weeks
* prior history of postpartum hemorrhage
* labor induction or augmentation with oxytocin
* advanced maternal age
* obesity with body mass index >40

Exclusion Criteria:

* a degree of case urgency to which taking time to consent for the study could compromise patient care, determined by anesthesiologist or obstetrician
* patient age <18 years or >50 years
* renal dysfunction with serum Creatinine > 1.0
* abnormal cardiac function or history of arrhythmia
* patient taking digoxin
* patient currently taking a calcium channel blocker for a cardiovascular indication

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study being conducted in pregnant women undergoing Cesarean delivery
Enrollment: 40 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh FRCA, Study Chair — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Investigators will consider sharing de-identified individual participant data including data analysis code with interested investigators on a case-by-case basis. Please email Dr. Ansari or Dr. Carvalho

REFERENCES:
- [Derived] Ansari JR, Kalariya N, Carvalho B, Flood P, Guo N, Riley E. Calcium chloride for the prevention of uterine atony during cesarean delivery: A pilot randomized controlled trial and pharmacokinetic study. J Clin Anesth. 2022 Sep;80:110796. doi: 10.1016/j.jclinane.2022.110796. Epub 2022 Apr 18. PMID 35447502

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium Chloride: Non-participating anesthesiologist prepares the drug solution, which is 1 gram of calcium chloride diluted into a total volume of 60 milliliters normal saline, labeled only with the study ID number. The solution is administered intravenously utilizing an Alaris syringe pump and microbore tubing, with infusion starting immediately at the time of fetal delivery at a rate of 360 milliliters per hour (for a calcium infusion rate of 100 milligrams /minute until the full 1 gram dose is administered).
  This is a one-time administration. Patients continue to receive all standard care during the Cesarean including 1 unit oxytocin bolus at the time of fetal delivery + continuous oxytocin infusion at 7.5 units per hour per our institution's protocol.
  Calcium Chloride: All included in intervention description.
  1 gram of calcium chloride in total 60 milliliters normal saline
- Placebo: Non-participating anesthesiologist prepares the placebo solution, which is 60 milliliters normal saline, labeled only with the study ID number. The solution is administered intravenously utilizing an Alaris syringe pump and microbore tubing, with infusion starting immediately at the time of fetal delivery at a rate of 360 milliliters per hour.
  This is a one-time administration. Patients continue to receive all standard care during the Cesarean including 1 unit oxytocin bolus at the time of fetal delivery + continuous oxytocin infusion at 7.5 units per hour per our institution's protocol.
  Placebo: 60 milliliters normal saline
Period: Overall Study
Arm/Group | Calcium Chloride | Placebo
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Chloride | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 4 | 6 | 10
  Race/Ethnicity: Black | 0 | 1 | 1
  Race/Ethnicity: Hispanic/Latina | 4 | 4 | 8
  Race/Ethnicity: White | 10 | 8 | 18
  Race/Ethnicity: Mixed | 1 | 1 | 2
  Race/Ethnicity: Other/Decline to disclose | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Gestational age [Median (Inter-Quartile Range); unit: weeks of gestation] | 38.4 [36.8 to 39.6] | 39.0 [35.7 to 39.7] | 38.6 [36.2 to 39.6]

OUTCOME MEASURES:

1. Primary Outcome: Uterine Atony
Description: The primary outcome of interest is the presence of clinical uterine atony, as defined the by any of the following:
  1. Administration of > 1 bolus of oxytocin
  2. Increase in the oxytocin infusion rate above the standard 7.5units/hour
  3. Administration of a second line uterotonic including methylergonovine, carboprost, or misoprostol
  4. Mechanical surgical interventions for uterine atony including placement of an intrauterine balloon, B-lynch sutures, or O'Leary sutures
  5. Requirement for embolization of the uterine arteries by interventional radiology
  6. Estimated blood loss> 1000 milliliters
  7. Transfusion of blood products during or within 4 hours of Cesarean
Time Frame: From time of fetal delivery until 4 hours after fetal delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 4 | 10

2. Secondary Outcome: Grading of Uterine Tone
Description: Subjective assessment of uterine tone by the obstetrician, from 0-100%.
  Obstetricians were blinded to study assignment arm, and were instructed that 0% indicates a completely atonic (un-contracted) uterus, and 100% indicates a perfectly, firmly contracted uterus. They were asked to provide this score by palpating the fundus (top) of the uterus as soon as the study drug infusion was complete.
Time Frame: A one-time value collected 10 minutes after Cesarean fetal delivery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 89 [80 to 90] | 80 [75 to 89]

3. Secondary Outcome: Estimated Blood Loss
Description: In milliliters. By blinded obstetrician, taking into account drape, sponge, and suction canister contents
Time Frame: Immediately upon surgery completion, as patient exits operating theater
Population: Quantitative blood loss was not able to be performed, so estimated blood loss was used for all participants
Measure: Median (Inter-Quartile Range); unit: milliters
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
milliters | 750 [600 to 800] | 850 [650 to 1000]

4. Secondary Outcome: Change in Hematocrit
Description: Changes from preoperative to standard postoperative day 1 hematocrit in patients. The hematocrit represents the percentage by volume of red blood cells in a blood sample and decreases after losing blood. The change in hematocrit was calculated by subtracting the number obtained the morning after surgery from the number obtained prior to surgery.
Time Frame: Drawn on postoperative day 1 as standard care
Measure: Mean (Standard Deviation); unit: hematocrit (%)
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
hematocrit (%) | 7.7 (4.4) | 6.7 (2.6)

5. Secondary Outcome: Total Crystalloid During Cesarean
Description: Amount of saline administered during cesarean
Time Frame: During entire Cesarean delivery record (generally about 2 hours)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
mL | 1200 [1000 to 2000] | 1750 [1500 to 2000]

6. Secondary Outcome: Maximum Increase in Heart Rate From Baseline (Beats Per Minute)
Description: Heart rate is recorded every minute throughout delivery. Heart rate values over the first 45 minutes after study drug completion will be compared to baseline calcium chloride to placebo group
Time Frame: first 45 minutes after study drug completion
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
beats per minute | 15.4 (8.8) | 14.2 (7.7)

7. Secondary Outcome: Maximal Decrease in Heartrate From Baseline
Description: Heart rate monitored for 45 minutes after study drug infusion (well past peak)
Time Frame: 45 minutes after study drug infusion is complete
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
beats per minute | 19.1 (13.1) | 16.7 (14.4)

8. Secondary Outcome: Maximal Increase in Mean Arterial Blood Pressure From Baseline
Description: Baseline mean arterial pressure was established upon entry into the operating room after at least 3 minutes had passed since positioning onto the operating room bed and prior to commencement of the cesarean delivery or to block placement. Mean arterial blood pressure was recorded every 5 minutes from this baseline timepoint until completion of the cesarean. Maximal increase was calculated as the difference between the baseline and the highest recorded mean arterial blood pressure.
Time Frame: While in the operating room, generally about 2 hours
Population: All participants
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
mmHg | 15.4 [11.0 to 19.8] | 14.2 [10.3 to 17.8]

9. Secondary Outcome: Maximal Decrease in Mean Arterial Blood Pressure From Baseline
Description: Baseline mean arterial pressure was established upon entry into the operating room after at least 3 minutes had passed since positioning onto the operating room bed and prior to commencement of the cesarean delivery or to block placement. Mean arterial blood pressure was recorded every 5 minutes from this baseline timepoint until completion of the cesarean. Maximal decrease was calculated as the difference between the baseline and the lowest recorded mean arterial blood pressure.
Time Frame: While in the operating room, generally about 2 hours
Population: All participants
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Calcium Chloride | Placebo
Number analyzed (Participants) | 20 | 20
mmHg | 33.8 [25.2 to 40.9] | 32.0 [21.1 to 43.7]

10. Secondary Outcome: Baseline Ionized Calcium Concentration
Description: Ionized calcium levels measured by phlebotomy. Analyzed prior to any study drug administration.
Time Frame: Prior to study drug (up to 5 minutes for blood draw)
Population: Because this outcome was assessed at baseline prior to study drug administration, participants in the active and placebo groups who consented to phlebotomy were combined for this analysis.
Measure: Mean (95% Confidence Interval); unit: millimol per liter
Groups:
- All Participants: All participants who consented to phlebotomy for ionized calcium level analysis
Arm/Group | All Participants
Number analyzed (Participants) | 24
millimol per liter | 1.18 [1.16 to 1.19]

11. Secondary Outcome: Clearance of Calcium Chloride
Description: Pharmacokinetic parameters were analyzed based upon ionized calcium concentrations over time. Blood calcium concentration was measured at the following time points: baseline (pre-drug delivery), 0-20 minutes after drug administration, and 20-90 minutes after delivery. The reported values for concentration over time were obtained using NONMEM (Non Linear Mixed Effects Modeling).
Time Frame: Samples drawn at baseline, at random time points after study drug administration while in the operating room, and upon arrival to the recovery room (up to 90 minutes)
Population: Patients who received calcium chloride and consented to blood sampling for PK analysis. Patients who received placebo were not included since they did not receive calcium chloride and had no data collected for the outcome.
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Calcium Chloride
Number analyzed (Participants) | 13
L/min | 0.93 [0.63 to 1.52]

12. Secondary Outcome: Volume of Distribution of Calcium Chloride
Description: Pharmacokinetic parameters were analyzed based upon ionized calcium concentrations over time. Blood calcium concentration was measured at the following time points: baseline (pre-drug delivery), 0-20 minutes after drug administration, and 20-90 minutes after delivery. The resulting values for concentration over time were evaluated with NONMEM
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Calcium Chloride
Number analyzed (Participants) | 13
Liters | 76 [49 to 91]

ADVERSE EVENTS:
Time Frame: Any event within the 5 days of delivery
Arm/Group | Calcium Chloride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Chloride (N=20) | Placebo (N=20)
IV line discomfort (Product Issues) | 1 (1) | 0 (0) — Mild changes in HR and blood pressure are defined as changes from the patient's baseline which are not associated with symptoms and did not require any treatment with medication or fluid.
Nausea or vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) — Any patient who experienced nausea or vomiting counted toward this tally.
Hypertension (Cardiac disorders) | 0 (0) | 2 (2) — Any hypertension above the patient's baseline blood pressure noted in the 30 minutes after starting study drug
Arrhythmia (Cardiac disorders) | 2 (2) | 3 (3) — Any bradycardia with heart rate <60, tachycardia with heart rate >100, or other arrhythmia (anything other than normal sinus rhythm) noted within 30 minutes of the study drug administration

LIMITATIONS AND CAVEATS:
This was a pilot study not designed to definitively assess primary and secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT03867383/Prot_SAP_001.pdf
  • Informed Consent Form (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT03867383/ICF_002.pdf